CLINICAL TRIAL: NCT03118557
Title: HLP-16-003H: Does a Twice Weekly, 12-week Pilates Pelvic Floor Strengthening Program Improve Short- and Long-term Measures of Stress Urinary Incontinence Symptoms in Women Ages 45-70 Years of Age.
Brief Title: Pilates Pelvic Floor Strengthening Program to Improve Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Deborah Rhodes, MD, Associate Professor of Medicine, College of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 17-001061
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Stress Urinary Incontinence
Keywords: pelvic floor; strengthening; Stress; urinary; incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilates pelvic floor strengthening exercise (Experimental)
  Interventions: Other: Pilates pelvic floor strengthening

INTERVENTIONS:
Other: Pilates pelvic floor strengthening — Pilates pelvic floor strengthening.

SUMMARY:
Does a twice weekly, 12-week Pilates pelvic floor strengthening program improve short- and long-term measures of stress urinary incontinence symptoms in women ages 45-70 years of age?

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-70 years of age.
2. Able to provide informed consent.
3. Able to lower and rise from the floor safely and independently.
4. Anticipated to be able to attend at least 9 of the first 12 classes (75%) in weeks 1-6.
5. Anticipated to be able to attend at least 9 of the final 12 classes (75%) in weeks 7-12.
6. Score of 6+ on ICIQ-UI Short Form.

Exclusion Criteria:

1. Pregnancy
2. Unable to speak and comprehend English
3. Chronic neurologic condition (e.g., Parkinson's or Multiple Sclerosis) that impacts bladder function.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Change in score on International Consultation on Incontinence (ICIQ-UI Short Form) | Baseline, 12 weeks
  The ICIQ-UI Short Form consists of 3 questions. The ICIQ score is a sum of the responses to the 3 questions with a total possible range of 0 (none) to 21 (all the time/a great deal).

SECONDARY OUTCOMES:
Change in score on Medical, Epidemiological, Social Aging (MESA) Urinary Incontinence Questionnaire | Baseline, 12 weeks
  The MESA Urinary Incontinence Questionnaire consists of 3 sections: General questions (unscored), Urge Incontinence (6 questions), and Stress Incontinence (9 questions). The scored questions can range from 0 (never) to 3 (often). The score for the Urge Incontinence is the sum of the responses/18, and the score for the Stress Incontinence section is the sum of the responses/27.
Change in score on Linear Analogue Self Assessment (LASA) | Baseline, 12 weeks
  The LASA questionnaire consists of 6 questions, each ranging from 0 (as bad as it can be) to 10 (as good as it can be). Therefore, the total possible scores would range from 0 (as bad as it can be) to 60 (as good as it can be).

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J Rhodes, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials